CLINICAL TRIAL: NCT03794752
Title: Evaluation of a Head Mounted Electronic Visual Enhancement Device in Low Vision Patients
Brief Title: Visual Enhancement Device in Low Vision Patients
Acronym: Evergaze
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Rafael Ufret-Vincenty, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU 012014-015
Record Dates: First submitted 2018-12-20; First posted 2019-01-07 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Macular Degeneration, Age-Related; Diabetic Retinopathy
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Participants will wear a head mounted visual enhancement device.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vision Aided by a Head Mounted Device (Other): A Head-Mounted Visual Enhancement Device developed by Evergaze Technology LLC has designed an electronic visual enhancement device that is compact and similar to glasses. It will be powered by a battery pack connected to the device. The electronic display will be affixed over only one of the user's eyes. The vision through the unobstructed eye will aid with the subject's balance and spatial orientation.
  Interventions: Device: Head-Mounted Visual Enhancement Device

INTERVENTIONS:
Device: Head-Mounted Visual Enhancement Device — Evergaze has designed a head mounted electronic visual enhancement device that is compact and similar to glasses. It is powered by a battery pack connected to the device. The electronic display will be affixed over only one of the participant's eye. The vision through the unobstructed eye will aid with the participant's balance and spatial orientation. The prototype display and camera will be connected to a battery pack/control box that will allow the user to quickly select one of 3 modes. Each mode will represent a combination of parameters (brightness of the display, focus lock, color/black & white, contrast, magnification) designed to optimize the image for different activities (e.g. reading, walking, computer use).

SUMMARY:
This study will be a prospective, non-randomized study of low-vision individuals diagnosed with either age-related macular degeneration (AMD) or diabetic macular edema with ETDRS visual acuity from 20/60 to 20/400 in both eyes from the University of Texas - Southwestern (UTSW) Medical Center at Dallas. Specifically, the primary objective of this testing is to establish the benefits of a wide field-of-view (FOV) monocular head-mounted visual enhancement device display (HMD), aiding the most degraded eye, as compared to best corrected visual acuity with glasses. It should be noted that in this approach, the HMD incorporates a camera, mounted coaxially with the visual axis of the eye with worse vision, and also image-enhancing or correction algorithms. Following review and execution of the informed consent, each subject will undergo an examination of their eyes, including: 1) ETDRS Best-corrected distance visual acuity; 2) Best-corrected near visual acuity; 3) Tests based on questions 5,6,7 and 11 of the National Eye Institute 25-item visual function questionnaire (NEI VFQ-25).

DETAILED DESCRIPTION:
A single visit, prospective, non-randomized study of low vision individuals diagnosed with Age Related Macular Degeneration or Diabetic macular edema research project is designed to last about 1.5 hours. All testing will be used for research purposes. There will be an 1) Early Treatment Diabetic Retinopathy Study visual acuity test, 2) near vision test, 3) Testing based on questions 5,6,7, and 11 of the National Eye Institute 25 item visual function questionnaire, (NEI VFQ-25) which includes a speed reading test, identifying objects, physically taking them and returning the items to correct original placement, once with glasses only, once with the head mounted visual device placed over the worst eye visually. There will also be an video tracks showing a conversation between 2 individuals - Subjects will be queried about the facial expressions of the actors during the conversation. The device is a wide field of view (FOV) monocular head-mounted visual enhancement device (HMD). The HMD has a camera mounted coaxially with the visual axis of the worse vision eye, and also image enhancing or correction algorithms. There are breaks planned between testing on the visual function exam portion of the NEI-25.

ELIGIBILITY:
Inclusion Criteria:

* Patient of any sex, race, or ethnicity who are 18 years of age or older. Spanish speaking patients will be encouraged to participate, Spanish forms will be available to review and execute.
* Patient willing to review, understand and sign written informed consent. Parents or legal guardians will consent on behalf of minors.
* Written authorization for use or release of health and research study information.
* Patient who volunteers is suffering from a posterior segment ophthalmic disorder including AMD and/or Diabetic Retinopathy and visual acuity from 20/60 to 20/400 in the better seeing eye.

Exclusion Criteria:

* Subjects will be excluded if they are less than 18 years of age.
* Subjects will not be considered for this research study if they will not review and execute the informed consent form.
* During the screening process, subjects will be excluded from further consideration if they are identified with having a potential ophthalmic diagnosis other than age-related macular degeneration or diabetic macular edema that could be negatively affecting the visual testing.
* ETDRS Visual Acuity better than 20/60 or worse than 20/400
* During screening, subjects will be disqualified from further assessment if it is determined that their refractive error is outside of the -5.00 to +5.00 D corrective range.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Ufret-Vincenty, MD, Principal Investigator — UTSW Medical Center

RESULTS

PARTICIPANT FLOW:
Groups:
- Use of Head Mounted Device: Evergaze has developed a head-mounted visual enhancement device for low-vision patients. Patients will be non-randomized individuals diagnosed with either Retinal Degeneration or diabetic macular edema with ETDRS (Early Treatment Diabetic Retinopathy Study) VA 20/60 to 20/400.
  The device will be placed over the most degraded eye incorporating a camera, mounted coaxially with the visual axis of the eye with the worse vision. Incorporation of a video recording of head and eye movement with the head mounted device is being included for any functionality improvements to be made. Then each subject will undergo complete examination of their eyes, including ETDRS VA, distance and near along with Questions 5,6,7,and 11 of the NEI (National Eye Institute) 25 item visual function questionnaire (NEI VFQ 25)
Period: Overall Study
Arm/Group | Use of Head Mounted Device
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants performing skills without the head mounted visual aid device will be provide the baseline values for each aspect of this study.
Arm/Group | Vision Aided by a Head Mounted Device
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Rows represent Race and Ethnicity.
  Participants
    Black | 1
    White/Hispanic | 1
    White/Non-HIspanic | 6

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity (BCVA) With the Head-mounted Electronic Visual Enhancement Device
Description: ETDRS chart will be used to assess best corrected visual acuity. The outcome with the participant using head-mounted electronic visual enhancement device.
  The single visit, prospective, non-randomized study of low vision individuals diagnosed with Age Related Macular Degeneration or Diabetic macular edema research project is designed to last about 1.5 hours.
Time Frame: 5 minutes post intervention
Measure: Count of Participants; unit: Participants
Groups:
- Vision Aided by a Head Mounted Device: ETDRS chart will be used to assess best corrected visual acuity. Change in best corrected visual acuity (BCVA) will be determined for each participant using the following conditions.
  1. The baseline with the participant not using head-mounted electronic visual enhancement device. 2. the outcome with the participant using head-mounted electronic visual enhancement device.
Arm/Group | Vision Aided by a Head Mounted Device
Number analyzed (Participants) | 8
Participants
  BCVA unable to read | 1
  BCVA </= 20/50 | 4
  BCVA </= 20/80 | 2
  BCVA > 20/350 | 1

2. Primary Outcome: Best Corrected Near Visual Acuity (BCNVA) With the Head-mounted Electronic Visual Enhancement Device
Description: ETDRS chart will be used to assess best corrected visual acuity. The outcome with the participant using head-mounted electronic visual enhancement device.
  A single visit, prospective, non-randomized study of low vision individuals diagnosed with Age Related Macular Degeneration or Diabetic macular edema research project is designed to last about 1.5 hours.
Time Frame: 10 minutes post intervention
Measure: Count of Participants; unit: Participants
Groups:
- Vision Aided by a Head Mounted Device: ETDRS chart will be used to assess best corrected visual acuity. Change in best corrected near visual acuity (BCNVA) will be determined for each participant using the following conditions.
  1. The baseline with the participant not using head-mounted electronic visual enhancement device. 2. the outcome with the participant using head-mounted electronic visual enhancement device.
Arm/Group | Vision Aided by a Head Mounted Device
Number analyzed (Participants) | 8
Participants
  BCVNA Unable to read | 1
  BCVNA <=20/50 | 2
  BCVNA <=20/150 | 1
  BCVNA > 20/150 | 4

3. Primary Outcome: Number of Participants Completing/Not Completing the Reading Assessments With the Head-mounted Electronic Visual Enhancement Device
Description: Reading completion with head-mounted electronic visual enhancement device was measured by reading a standard paragraph from 3-Minute Reading Assessments by Rasinski TV and Padak N, 2005. Scholastic Inc., NY.
Time Frame: Day 1 up to 6 minutes post intervention
Population: Participants were asked to read a passage 98 words within a 3 min. time period
Measure: Count of Participants; unit: Participants
Groups:
- Vision Aided by a Head Mounted Device: Reading speed is measured by using a standard paragraph. English Paragraph Reference: 3-Minute Reading Assessments, Rasinski TV and Padak N, 2005. Scholastic Inc., NY.
  This outcome examines change in reading speed of the participant in two separate conditions:
  1. Baseline reading - no use of the head-mounted electronic visual enhancement device. and 2. reading using head-mounted electronic visual enhancement device.
Arm/Group | Vision Aided by a Head Mounted Device
Number analyzed (Participants) | 8
Participants
  Completed reading assignment with device | 4
  Did not complete reading assignment with device | 4

4. Primary Outcome: Number of Participants Able/Unable to Identify Facial Expressions With the Head-mounted Electronic Visual Enhancement Device.
Description: Face sheet and video are shown to the subject to identify facial expression and time taken is recorded. Change in response speed to identify facial expressions using the head-mounted electronic visual enhancement device.
  A single visit, prospective, non-randomized study of low vision individuals diagnosed with Age Related Macular Degeneration or Diabetic macular edema research project is designed to last about 1.5 hours.
Time Frame: Day 1 up to 1 minute post intervention
Measure: Count of Participants; unit: Participants
Groups:
- Vision Aided by a Head Mounted Device: Face sheet and video are shown to the subject to identify facial expression and time taken is recorded. Change in response speed to identify facial expressions will be determined for each participant using the following conditions.
  1. Using the head-mounted electronic visual enhancement device. 2. Without using the head-mounted electronic visual enhancement device.
Arm/Group | Vision Aided by a Head Mounted Device
Number analyzed (Participants) | 8
Participants
  Able to distinguish expressions w/ device | 4
  Unable to distinguish expressions w/ device | 4

5. Primary Outcome: Response Speed to Visual-motor Skills to Identify Shapes and Objects With the Head-mounted Electronic Visual Enhancement Device
Description: Portable shelf storage is placed at 5-feet distance and time taken to identify shapes and objects is recorded with the head-mounted electronic visual enhancement device.
  A single visit, prospective, non-randomized study of low vision individuals diagnosed with Age Related Macular Degeneration or Diabetic macular edema research project is designed to last about 1.5 hours.
Time Frame: Initial Baseline and 3 minutes
Measure: Count of Participants; unit: Participants
Groups:
- Vision Aided by a Head Mounted Device: Portable shelf storage is placed at 5-feet distance and time taken to identify shapes and objects is recorded. Data will record change in response speed to identify shapes and objects under 2 conditions; 1. with the participant using the head-mounted electronic visual enhancement device and 2. with the participant not using the head-mounted electronic visual enhancement device .
Arm/Group | Vision Aided by a Head Mounted Device
Number analyzed (Participants) | 8
Participants
  Identify items with device < 15 sec w/ headset | 3
  Identify items with device > 15 sec w/ headset | 3
  Cannot identify items w/ headset | 2

ADVERSE EVENTS:
Time Frame: A single visit, prospective, non-randomized study of low vision individuals diagnosed with Age Related Macular Degeneration or Diabetic macular edema research project is designed to last about 1.5 hours.
Arm/Group | Use of Head Mounted Device
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
This study had a small enrollment of 8 initial pilot study participants that were tested but not analyzed due to an early termination of the study. Termination was due to irreconcilable differences regarding intellectual property.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT03794752/Prot_SAP_000.pdf